CLINICAL TRIAL: NCT04001556
Title: RElevance of UltraSonography for Assessing Salivary Gland Involvement in Systemic Sclerosis (SSc)
Acronym: REUSSI-SSc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 35RC18_9905
Record Dates: First submitted 2019-04-01; First posted 2019-06-28 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: cross-sectionnal pilot study
Who Masked: Outcomes Assessor
Masking Description: The examiner performin the evaluation of ultrasound features of the main salivary glands will not have acess at the first part of patient evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients reporting subjective sicca symptoms (Experimental): HAQ(Health Assessment Questionnaire) Score, bilateral schirmer 's test, unstimulated whole salivary flow rate, blood sample for immunologic evaluation
  Interventions: Diagnostic Test: Minor Salivary gland Biopsy; Diagnostic Test: ARFI; Diagnostic Test: MSG US
- Patients without subjective sicca symptoms (Experimental): HAQ(Health Assessment Questionnaire) score, bilateral schirmer 's test, unstimulated whole salivary flow rate, blood sample for immunologic evaluation
  Interventions: Diagnostic Test: ARFI; Diagnostic Test: MSG US

INTERVENTIONS:
Diagnostic Test: Minor Salivary gland Biopsy — Minor salivary gland biopsy with injection of lidocain
  Arms: Patients reporting subjective sicca symptoms
Diagnostic Test: ARFI — Acoustic Radiation Force Impulse on Major Salivary Glands
Diagnostic Test: MSG US — Ultrasonography of Major Salivary Glands

SUMMARY:
As fibrosis of salivary glands is supposed to be the main mechanism involved in Systemic sclerosis (SSc)-associated sicca syndrome, Ultrasonography , biopsy and measuring gland elasticity (by ARFI (Acoustic Radiation Force Impulse)) in SSc patients could also constitute a relevant method to assess the potential alterations of echostructure of major salivary glands and the fibrosis of Salivary Glands in this disease.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a rare autoimmune chronic disorder characterised by vascular hyper-reactivity and fibrosis of the skin as well as internal organs. Intimal hyperplasia, endothelial dysfunction and occlusive vasculopathy are the underlying basis of these chronic vascular damages. The expression of the vasculopathy especially includes Raynaud phenomenon (RP), digital ulcers (DUs), gastro-intestinal involvement and pulmonary arterial hypertension (PAH). Sicca syndrome is clinically characterised by dryness of the eyes (xerophthalmia) and mouth (xerostomia). The prevalence of sicca symptoms is up to 70% in prospective series of SSc patients. Sicca syndrome is supposed to be primarily related to glandular fibrosis. The prevalence of primary Sjögren Syndrome (pSS) among SSc patients, as defined by the American-European Consensus Group criteria is around 15%. Sicca syndrome is therefore a frequent feature in SSc and constitutes an important cause of quality of life's impairment in SSc If studies have already evaluated clinical and histological alterations of minor salivary glands secondary to sicca syndrome in SSc , only few studies used the recent ACR(American College of Rheumatology) 2013 classification criteria for SSc to select patients. SGUS(Salivary Gland UltraSonography) evaluation in SSc has never been assessed to date. Potential alterations of MSG (Major Salivary Gland) echostructure in SSc have never been described to date. The performances and reliability of SGUS to assessed MSG involvement in SSc are still to be determined. As fibrosis of salivary glands is supposed to be the main mechanism involved in SSc-associated sicca syndrome, measuring salivary-gland elasticity using ARFI-ultrasonography in SSc patients could also constitute a relevant method to assess the fibrosis of MSG in this disease. A cross-sectional pilot study is therefore needed to explore these relevant questions about sicca syndrome in SSc.

ELIGIBILITY:
Inclusion Criteria:

* Patients over eighteen years old;
* Fulfilling 2013 ACR classification criteria for Systemic sclerosis (Van den Hoogen et al. 2013);
* 60 patients with subjective sicca symptoms reported by a standardised questionnaire (Vitali C et al. 2002);
* 15 patients without sicca symptoms;
* Who has signed an informed consent
* Benefiting from a social security scheme

Exclusion Criteria:

* Treatment: current (or in the past 6 months) immunosuppressive treatment by rituximab or cyclophosphamide (representing less than 5% of SSc patients in the investigator's centres);
* Current (or in the past 6 months) treatment with drugs with anti-cholinergic properties (Selective Serotonin Reuptake Inhibitors and anti-histaminic inhibitors (hydroxyzine));
* Current treatment with antiplatelet aggregates
* Anti-vitamin K treatment (increasing risk of bleeding during minor salivary gland biopsy); and oral anti-coagulant
* Known abnormal coagulation (prolonged aPPT(activated partial thromboplastin time) and / or PT (Prothrombin time ( <70%)), or known thrombocytopenia (<150,000 platelets / mm3)
* Known secondary sicca symptoms : history of head-and-neck radiotherapy, hepatitis C infection, AIDS, sarcoidosis, amyloidosis, graft-vs-host disease and IgG4(Isotype's immunoGlobulin G4)-related disease;
* Pregnancy or breastfeeding mothers;
* Known intolerance/allergy to xylocain injection;
* Adults legally protected (under judicial protection, guardianship, or supervision), inability to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Ultrasonography characteristics of major salivary glands | up to six months (at evaluation visit)
  Ultrasonography characteristics of major salivary glands based on Salaffi's composite score.
  each MSG will be scored as followed:
  * grade 0 = normal homogeneous glands;
  * grade 1 = Homogenous borders, slightly heterogeneous parenchyma,
  * grade 2 = Homogenous borders, multiple hypoechogenic areas measuring < 2 mm,
  * grade 3 = multiple hypoechogenic areas measuring 2-6 mm or irregular borders or invisible posterior part of the gland;
  * grade 4 = unstructured glandular parenchyma with multiple hypoechogenic areas measuring >6 mm or calcifications with echogenic bands.
  In each patient, 4 grades can be obtained (1 grade per gland);
  the sum of these 4 grades (range 0-16) will be the Salaffi's score.
  A score of 0 has the best outcome, of 16 the worse
Ultrasonography characteristics of major salivary glands | up to six months (at evaluation visit)
  Ultrasonography characteristics of major salivary glands based on bilateral ARFI(Acoustic radiation force Impulse) elastometry

SECONDARY OUTCOMES:
Variants of the Salaffi score | up to six months (evaluation visit)
  Scores of Hocevar,based on the same ultrasound parameters but with a weighting different from that of Salaffi in the calculation of the score.
  Echostructure of the four salivary glands will be graded 0 to 12 ; the sum of these 4 grades (range 0-48) will be the Hocevar's score. A score of 0 has the best outcome, of 48 the worse.
Variants of the Salaffi score | up to six months (evaluation visit)
  Scores of Milic,based on the same ultrasound parameters but with a weighting different from that of Salaffi in the calculation of the score.
  Echostructure of the four salivary glands will be graded 0 to 3 ; the sum of these 4 grades (range 0-12) will be the Milic's score. A score of 0 has the best outcome, of 12 the worse.
Variants of the Salaffi score | up to six months (evaluation visit)
  Scores Jousse-Joulin / Cornec constituting , based on the same ultrasound parameters but with a weighting different from that of Salaffi in the calculation of the score.
  Echostructure of the four salivary glands will be graded 0 to 4 ; the sum of these 4 grades (range 0-16) will be the Jousse-Joulin/Cornec's score.
  A score of 0 has the best outcome, of 16 the worse.
Biopsy of the minor salivary glands | up to six months (evaluation visit)
  Biopsies of the minor salivary glands with standardized histological characterization of the Chisholm score.
  Chisholm'score will evaluate the number of lymphocytic foci/4mm2 grade 1 : none or slight, grade 2 : less than 50 lymphocytes and histocytes, grade 3 : one focus with at least 50 lymphocytes, grade 4 : More than one focus with at least 50 lymphocytes,
  Grade 1 has the best outcome, grade 4 the worse.
Biopsy of the minor salivary glands | up to six months (evaluation visit)
  Biopsies of the minor salivary glands with standardized characterization of the focus score.
  Focus score : the number of mononuclear cell infiltrates containing at least 50 inflammatory cells in a 4 mm2 glandular section,
  Focus score 0 = no mononuclear cell infiltrate containing at least 50 inflammatory cells in a 4 mm2 glandular section,
  Focus score =1 or >1 : one or more mononuclear cell infiltrates containing at least 50 inflammatory cells in a 4 mm2 glandular section,
  Focus score 0 has the best outcome Focus score =1 or >1 has the worse outcome
Biopsy of the minor salivary glands | up to six months (evaluation visit)
  Biopsies of the minor salivary glands with evaluation of fibrosis assessed from F1 to F4
Evaluation of the presence or absence of objective criteria of Sjogren | up to six months (evaluation visit)
  Evaluation of the presence or absence of objective criteria of Sjogren according to salivary flow test
Evaluation of the presence or absence of objective criteria of Sjogren | up to six months (evaluation visit)
  Evaluation of the presence or absence of objective criteria of Sjogren according to Schirmer test.
Clinical evaluation of systemic scleroderma lesions | up to six months (evaluation visit)
  forms of the disease
Clinical evaluation of systemic scleroderma lesions | up to six months (evaluation visit)
  duration of evolution of the disease
Clinical evaluation of systemic scleroderma lesions | up to six months (evaluation visit)
  visceral damage : Presence or absence of pulmonary involvement on CT scan, Presence or absence of pulmonary arterial hypertension on echocardiography.
Clinical evaluation of systemic scleroderma lesions | up to six months (evaluation visit)
  immunological data : Positivity of : Anti SSA(Anti Sjögren Syndrom A) antibodies,Anti SSb(Anti Sjögren syndrom B) antibodies,Anti Topoisomerase antibodies, Anti Centromere antibodies, Anti RNA polymerase III antibodies
  Using Indirect ImmunoFluorescence (IFI) ( as binary parameter (positive or negative)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick JEGO, MD, Principal Investigator — University Hospital of Rennes
Locations (3):
- France (3):
  - CHU Brest Service de Rhumatologie, Brest
  - CHU rennes, Rennes
  - CHU Tours, Service de médecine interne, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salaffi F, Argalia G, Carotti M, Giannini FB, Palombi C. Salivary gland ultrasonography in the evaluation of primary Sjogren's syndrome. Comparison with minor salivary gland biopsy. J Rheumatol. 2000 May;27(5):1229-36. PMID 10813292
- [Background] Hocevar A, Ambrozic A, Rozman B, Kveder T, Tomsic M. Ultrasonographic changes of major salivary glands in primary Sjogren's syndrome. Diagnostic value of a novel scoring system. Rheumatology (Oxford). 2005 Jun;44(6):768-72. doi: 10.1093/rheumatology/keh588. Epub 2005 Mar 1. PMID 15741192
- [Background] Milic VD, Petrovic RR, Boricic IV, Radunovic GL, Pejnovic NN, Soldatovic I, Damjanov NS. Major salivary gland sonography in Sjogren's syndrome: diagnostic value of a novel ultrasonography score (0-12) for parenchymal inhomogeneity. Scand J Rheumatol. 2010 Mar;39(2):160-6. doi: 10.3109/03009740903270623. PMID 20059370
- [Background] Jousse-Joulin S, Milic V, Jonsson MV, Plagou A, Theander E, Luciano N, Rachele P, Baldini C, Bootsma H, Vissink A, Hocevar A, De Vita S, Tzioufas AG, Alavi Z, Bowman SJ, Devauchelle-Pensec V; US-pSS Study Group. Is salivary gland ultrasonography a useful tool in Sjogren's syndrome? A systematic review. Rheumatology (Oxford). 2016 May;55(5):789-800. doi: 10.1093/rheumatology/kev385. Epub 2015 Dec 14. PMID 26667216
- [Background] Cornec D, Jousse-Joulin S, Pers JO, Marhadour T, Cochener B, Boisrame-Gastrin S, Nowak E, Youinou P, Saraux A, Devauchelle-Pensec V. Contribution of salivary gland ultrasonography to the diagnosis of Sjogren's syndrome: toward new diagnostic criteria? Arthritis Rheum. 2013 Jan;65(1):216-25. doi: 10.1002/art.37698. PMID 23108632